CLINICAL TRIAL: NCT00627796
Title: A Multicenter, Open, Prospective, Observational Study to Investigate the Effect of Lanreotide Autogel 120 mg on Control of GH and IGF-I Excess and Tumor Shrinkage in Newly Diagnosed Patients With Acromegaly
Brief Title: Lanreotide Autogel-120 mg as First-Line Treatment of Acromegaly
Acronym: ATG1line
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Genova (Other)
Responsible Party: Annamaria Colao, University Federico II
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-9
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2007-12

CONDITIONS: Acromegaly
Keywords: GH; IGF-I; tumor; lanreotide
MeSH Terms: conditions — Acromegaly; Neoplasms | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Newly diagnosed patients with acromegaly
  Interventions: Drug: Lanreotide-Autogel 120 mg

INTERVENTIONS:
Drug: Lanreotide-Autogel 120 mg — ATG120 mg is given as deep subcutaneous injection into the buttock. Each patient receives one deep subcutaneous injection of ATG120 mg at Visit 1 (V1) and subsequent injection every 4 weeks for 3 injections. Based on GH levels, the dosing interval has been determined as follows: if GH levels were > 2.5 mcg/l, ATG 120 mg is given every 4 weeks while if they were < 2.5 mcg/l ATG 120 mg is administered every 6 weeks for another 3 injections. Afterwards, the dose is maintained as above except in patients with GH levels <1 mcg/l receiving ATG 120 mg every 8 weeks. The estimated duration of treatment is 48-52 weeks according with dose titration.
  Other Names: Ipstyl

SUMMARY:
Recently, a new formulation of lanreotide, lanreotide Autogel (ATG) 60 mg, 90 mg and 120 mg was developed in order to further extend the duration of the release of the active ingredient. The ATG formulation consists of a solution of lanreotide in water with no additional excipients. ATG was found to have linear pharmacokinetics for the 60 to 120 mg doses and provided a prolonged dosing interval and good tolerability (1). In some previous studies, the ATG was demonstrated as effective as the micro-particle lanreotide (2,3) and as octreotide-LAR in patients with acromegaly (4-7).

Data on the efficacy of ATG in newly diagnosed patients with acromegaly are still lacking. Similarly, the prevalence and amount of tumor shrinkage after ATG treatment is unknown. This information is particularly useful in the setting of first-line therapy of acromegaly that is currently becoming a more frequent approach to the disease (8). It is demonstrated that approximately 80% of the patients treated with depot somatostatin analogues as first line have a greater than 20% tumor shrinkage during the first 12 months of treatment (9). A definition of significant tumor shrinkage was provided in 14 studies (including a total number of patients of 424) and the results showed that 36.6% (weighted mean percentage) of patients receiving first-line somatostatin analogues therapy for acromegaly had a significant reduction in tumor size (10). About 50% of the patients were found to have a greater than 50% tumor shrinkage within the first year of treatment (10); in this study we found that percent decrease in IGF-I levels was the major determinant of tumor shrinkage (10).

The current open, prospective study is designed to investigate the prevalence and amount of tumor shrinkage in newly diagnosed patients with acromegaly treated first-line with ATG.

DETAILED DESCRIPTION:
This is an open, prospective, observational, clinical study to be performed in two University Hospitals (Naples and Genova, Italy). The primary objective is to evaluate the efficacy of the ATG 120 mg on control of GH and IGF-I excess in acromegaly according with the currently accepted criteria (12) and on tumor shrinkage. The secondary objectives are to assess improvement of clinical symptoms and safety profile. The study population will consist of at least 20 patients, enrolled in the two centers from Jan 1st 2003 to June 30th 2007. Patients give their written informed consent prior to entering into the study. The study was performed according to the principles defined by the declaration The safety population, as defined by the protocol, consists of patients who received at least one study drug dosing.

Hormonal evaluation GH levels are assessed as a mean value of 5 samples at 30-min intervals (starting between 08:00 and 9:00 in the morning) taken at each visit before the injection of ATG. IGF-I levels are assessed as a single sample taken at each visit at the same time as the first GH sample. All hormonal parameters were assessed in a central laboratory (University of Genoa).

Improvement in clinical symptoms is considered on the basis of a semiquantitative scale for asthenia, hyperhidrosis, headache, swelling of extremities, arthralgia, paraesthesia, carpal tunnel syndrome: symptoms were graded as 0 = absent, 1 = mild, 2 = moderate, 3 = severe.

Any adverse event (AE) during the study is monitored and reported by the investigators. Safety, evaluated by local laboratory data, is assessed at inclusion and at the final visit by: hematology: erythrocytes, leukocytes, platelets, haemoglobin, hematocrit; biochemistry: glucose, creatinine, alkaline phosphatase, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), electrolytes (sodium, potassium, calcium, phosphorous) glycosylated haemoglobin, triglycerides, total and high density lipoproteins (HDL) cholesterol, blood amylase, iron, transferrin, prothrombin; glucose and insulin concentrations; hormonal evaluation: thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), free triiodothyronine (FT4), follicle stimulating hormone (FSH) and luteinizing hormone (LH) levels. Safety related to gallbladder is assessed by ultrasound examination performed at inclusion and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active acromegaly [serum GH levels above 2.5 μg/liter and/or above 1 μg/liter after oral glucose tolerance test (OGTT) and abnormal IGF-I values] with a micro- (<10 mm max tumor diameter) or macroadenoma (>10 mm max tumor diameter)
* Patients never treated before
* Patients who do not require immediate surgery because of neurological symptoms and/or emergency conditions
* Patients who signed an informed consent to participate to the study.

Exclusion Criteria:

* Patients already treated before with surgery or radiotherapy or with medical treatment
* Patients with mixed GH-PRL adenomas who require combined somatostatin and dopamine treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Control of GH and IGF-I excess and tumor shrinkage | 3 and 12 months

SECONDARY OUTCOMES:
Improvement of clinical symptoms and safety profile | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- Annamaria Colao, Naples, Italy

REFERENCES:
- [Result] Antonijoan RM, Barbanoj MJ, Cordero JA, Peraire C, Obach R, Valles J, Cherif-Cheikh R, Torres ML, Bismuth F, Montes M. Pharmacokinetics of a new Autogel formulation of the somatostatin analogue lanreotide after a single subcutaneous dose in healthy volunteers. J Pharm Pharmacol. 2004 Apr;56(4):471-6. doi: 10.1211/0022357023123. PMID 15099442
- [Result] Caron P, Beckers A, Cullen DR, Goth MI, Gutt B, Laurberg P, Pico AM, Valimaki M, Zgliczynski W. Efficacy of the new long-acting formulation of lanreotide (lanreotide Autogel) in the management of acromegaly. J Clin Endocrinol Metab. 2002 Jan;87(1):99-104. doi: 10.1210/jcem.87.1.8153. PMID 11788630
- [Result] Lucas T, Astorga R; Spanish-Portuguese Multicentre Autogel Study Group on Acromegaly. Efficacy of lanreotide Autogel administered every 4-8 weeks in patients with acromegaly previously responsive to lanreotide microparticles 30 mg: a phase III trial. Clin Endocrinol (Oxf). 2006 Sep;65(3):320-6. doi: 10.1111/j.1365-2265.2006.02595.x. PMID 16918950
- [Result] Ashwell SG, Bevan JS, Edwards OM, Harris MM, Holmes C, Middleton MA, James RA. The efficacy and safety of lanreotide Autogel in patients with acromegaly previously treated with octreotide LAR. Eur J Endocrinol. 2004 Apr;150(4):473-80. doi: 10.1530/eje.0.1500473. PMID 15080776
- [Result] Alexopoulou O, Abrams P, Verhelst J, Poppe K, Velkeniers B, Abs R, Maiter D. Efficacy and tolerability of lanreotide Autogel therapy in acromegalic patients previously treated with octreotide LAR. Eur J Endocrinol. 2004 Sep;151(3):317-24. doi: 10.1530/eje.0.1510317. PMID 15362960
- [Result] van Thiel SW, Romijn JA, Biermasz NR, Ballieux BE, Frolich M, Smit JW, Corssmit EP, Roelfsema F, Pereira AM. Octreotide long-acting repeatable and lanreotide Autogel are equally effective in controlling growth hormone secretion in acromegalic patients. Eur J Endocrinol. 2004 Apr;150(4):489-95. doi: 10.1530/eje.0.1500489. PMID 15080778
- [Result] Ronchi CL, Boschetti M, Degli Uberti EC, Mariotti S, Grottoli S, Loli P, Lombardi G, Tamburrano G, Arvigo M, Angeletti G, Boscani PF, Beck-Peccoz P, Arosio M; Italian Multicenter Autogel Study Group in Acromegaly. Efficacy of a slow-release formulation of lanreotide (Autogel) 120 mg) in patients with acromegaly previously treated with octreotide long acting release (LAR): an open, multicentre longitudinal study. Clin Endocrinol (Oxf). 2007 Oct;67(4):512-9. doi: 10.1111/j.1365-2265.2007.02917.x. Epub 2007 Jun 7. PMID 17555511
- [Result] Colao A, Martino E, Cappabianca P, Cozzi R, Scanarini M, Ghigo E; A.L.I.C.E. Study Group. First-line therapy of acromegaly: a statement of the A.L.I.C.E. (Acromegaly primary medical treatment Learning and Improvement with Continuous Medical Education) Study Group. J Endocrinol Invest. 2006 Dec;29(11):1017-20. doi: 10.1007/BF03349217. No abstract available. PMID 17259801
- [Result] Bevan JS. Clinical review: The antitumoral effects of somatostatin analog therapy in acromegaly. J Clin Endocrinol Metab. 2005 Mar;90(3):1856-63. doi: 10.1210/jc.2004-1093. Epub 2004 Dec 21. PMID 15613435
- [Result] Melmed S, Sternberg R, Cook D, Klibanski A, Chanson P, Bonert V, Vance ML, Rhew D, Kleinberg D, Barkan A. A critical analysis of pituitary tumor shrinkage during primary medical therapy in acromegaly. J Clin Endocrinol Metab. 2005 Jul;90(7):4405-10. doi: 10.1210/jc.2004-2466. Epub 2005 Apr 12. PMID 15827109
- [Derived] Colao A, Auriemma RS, Rebora A, Galdiero M, Resmini E, Minuto F, Lombardi G, Pivonello R, Ferone D. Significant tumour shrinkage after 12 months of lanreotide Autogel-120 mg treatment given first-line in acromegaly. Clin Endocrinol (Oxf). 2009 Aug;71(2):237-45. doi: 10.1111/j.1365-2265.2008.03503.x. Epub 2008 Dec 15. PMID 19094074